CLINICAL TRIAL: NCT06145022
Title: Effect of a Stress Reduction and Lifestyle Modification Programme on the Quality of Life of Irritable Bowel Syndrome Patients (MBM IBS)
Brief Title: Stress Reduction and Lifestyle Modification in Irritable Bowel Syndrome Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Bavarian State Ministry of Health and Care (Other Government)
Responsible Party: Principal Investigator, Jost Langhorst, Prof. Dr. med., Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23065
Record Dates: First submitted 2023-11-10; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: lifestyle modification; Mind-Body medicine; integrative medicine
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Once a week for 10 weeks with a circumference of 60 hours with mindfulness-based stress reduction and further process of the Mind / body medicine.
  Interventions: Behavioral: lifestyle modification
- waitlist control group (Active Comparator): A unique education unit within the scope of 1,5 hours on the influence of lifestyle factors on the disease and self-help materials for the independent training. After the follow-up measurement opportunity to participate in the program.
  Interventions: Behavioral: waitlist control group

INTERVENTIONS:
Behavioral: lifestyle modification — The group intervention is carried out once a week for 10 weeks for a total of 60 hours with elements of mindfulness-based stress reduction (MBSR) and mind / body medicine. In this project, this program will be adapted to the specific needs of irritable bowel syndrome patients.
  Arms: intervention group
Behavioral: waitlist control group — Participants in this group receive a one-time education unit within the scope of 1,5 hours on the influence of lifestyle factors on the disease, also self-help materials for independent training offered. Following the follow-up measure also this group is given the opportunity to participate in the multimodal stress reduction- and lifestyle modification program.
  Arms: waitlist control group

SUMMARY:
In the planned efficacy study, a prospective randomized controlled trial will be conducted to investigate the extent to which a multimodal stress reduction and lifestyle modification program can be reflected in patients with irritable bowel syndrome (IBS) within the framework of a clinical study. For this purpose, 118 patients with IBS will be enrolled in a clinical study. The intervention group will participate in a partial outpatient multimodal stress reduction and lifestyle modification program over 10 weeks, while the waitlist control group will only receive an educational session and written information on treatment and self-help options. The primary research question encompasses the examination of the program's impact on the severity of symptoms associated with irritable bowel syndrome (measured with the IBS-Symptom Severity Scale [IBS-SSS]) and additionally its influence on quality of life, stress, and mental well-being. Another aspect of the study is the utilization of medical services (e.g., comparing the number of doctor visits; intake of prescribed and over-the-counter medications). Additionally, a comparison of days of work disability will be conducted.

DETAILED DESCRIPTION:
The intervention is a 10-week multimodal stress reduction and lifestyle modification program consisting of 10 sessions, each lasting 6 hours. In groups of around 10 individuals, patients are comprehensively trained on the interplay between lifestyle and health, stress management, moderate physical activity (including yoga and Tai Chi), a Mediterranean diet, and self-help strategies. Successfully tested in two pilot studies, the program has evolved over 15 years and gained clinical experience in chronic inflammatory bowel diseases. It is now being applied to patients with irritable bowel syndrome (IBS).

Built on concepts like the Mind-Body Program and mindfulness-based stress reduction, the intervention incorporates elements from salutogenic and transtheoretical models and psychotherapeutic approaches.

Few integrative medicine approaches for IBS have undergone rigorous evaluation. IBS patients often experience reduced quality of life due to stress and psychosocial symptoms. The program, proven effective in inflammatory bowel diseases, covers stress reduction, dietary improvement, physical activity promotion, self-care applications, coping strategy training, and naturopathic treatments. Medically supervised, the group setting aims to enhance the intervention's impact through mutual support. Practical skills are demonstrated, and the goal is to empower patients for active, responsible, long-term management.

Participants in the waitlist control group receive a 1,5-hour educational session on lifestyle factors' influence and self-help materials. After week 36 measurements, they are offered participation in the multimodal program.

Questionnaires, a diary, and interviews will measure the outcomes of the study. Sociodemographics will be collected.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of irritable bowel syndrome (IBS with diarrhea, IBS with constipation, mixed-type IBS, or unspecified IBS); IBS-SSS Score > 75

Exclusion Criteria:

* Severe mental illness (e.g., clinically significant depression, substance use disorder, schizophrenia)
* Severe comorbid somatic illness (e.g., oncological disease)
* Pregnancy
* Participation in other stress reduction programs or clinical studies on psychological interventions
* Known intolerances (fructose, lactose), celiac disease, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Severity of IBS symptoms by IBS-SSS | week 0
  Irritable bowel syndrome severity scoring system (IBS-SSS); 5-item questionnaire; scale from 0% (= not at all) to 100% (= very severe); cut-off of IBS-SSS scores to evaluate the severity of IBS: < 175 for mild IBS, 175-300 for moderate IBS, and > 300 for severe IBS
Severity of IBS symptoms by IBS-SSS | week 12
  Irritable bowel syndrome severity scoring system (IBS-SSS); 5-item questionnaire; scale from 0% (= not at all) to 100% (= very severe); cut-off of IBS-SSS scores to evaluate the severity of IBS: < 175 for mild IBS, 175-300 for moderate IBS, and > 300 for severe IBS
Severity of IBS symptoms by IBS-SSS | week 36
  Irritable bowel syndrome severity scoring system (IBS-SSS); 5-item questionnaire; scale from 0% (= not at all) to 100% (= very severe); cut-off of IBS-SSS scores to evaluate the severity of IBS: < 175 for mild IBS, 175-300 for moderate IBS, and > 300 for severe IBS
overall change in health status | week 12
  Rating scale from 1 (= much worse) to 5 (= much better)
overall change in health status | week 36
  Rating scale from 1 (= much worse) to 5 (= much better)

SECONDARY OUTCOMES:
Disease related Quality of Life by IBS-QOL | week 0
  The IBS-QOL is a self-report quality-of-life measure specific to Irritable Bowel Syndrome (IBS) that can be used to assess the impact of IBS and its treatment. 34 items with a 5-point response scale from 1 (=not at all) to 5 (= Extremely/a great deal); 34 items are summed and averaged for a total score and then transformed to a 0-100 scale for ease of interpretation with higher scores indicating better IBS specific quality of life.
Disease related Quality of Life by IBS-QOL | week 12
  The IBS-QOL is a self-report quality-of-life measure specific to Irritable Bowel Syndrome (IBS) that can be used to assess the impact of IBS and its treatment. 34 items with a 5-point response scale from 1 (=not at all) to 5 (= Extremely/a great deal); 34 items are summed and averaged for a total score and then transformed to a 0-100 scale for ease of interpretation with higher scores indicating better IBS specific quality of life.
Disease related Quality of Life by IBS-QOL | week 36
  The IBS-QOL is a self-report quality-of-life measure specific to Irritable Bowel Syndrome (IBS) that can be used to assess the impact of IBS and its treatment. 34 items with a 5-point response scale from 1 (=not at all) to 5 (= Extremely/a great deal); 34 items are summed and averaged for a total score and then transformed to a 0-100 scale for ease of interpretation with higher scores indicating better IBS specific quality of life.
General Quality of Life by EQ-5D-SL | week 0
  The EQ-5D assesses health status in terms of five dimensions of health (mobility, self-care, usual activities, pain and discomfort, and anxiety and depression) and is considered a 'generic' questionnaire because these dimensions are not specific to any one patient group or health condition. 5-point response-scale from 1 (=not /no problems) to 5 (=unable to [mobility, self-care, usual activities]/extreme [pain/depression]/extremely [anxiety/depression]); result: 5-digit health status profile that represents that person's level of reported problems on the five EQ-5D health dimensions
General Quality of Life by EQ-5D-SL | week 12
  The EQ-5D assesses health status in terms of five dimensions of health (mobility, self-care, usual activities, pain and discomfort, and anxiety and depression) and is considered a 'generic' questionnaire because these dimensions are not specific to any one patient group or health condition. 5-point response-scale from 1 (=not /no problems) to 5 (=unable to [mobility, self-care, usual activities]/extreme [pain/depression]/extremely [anxiety/depression]); result: 5-digit health status profile that represents that person's level of reported problems on the five EQ-5D health dimensions
General Quality of Life by EQ-5D-SL | week 36
  The EQ-5D assesses health status in terms of five dimensions of health (mobility, self-care, usual activities, pain and discomfort, and anxiety and depression) and is considered a 'generic' questionnaire because these dimensions are not specific to any one patient group or health condition. 5-point response-scale from 1 (=not /no problems) to 5 (=unable to [mobility, self-care, usual activities]/extreme [pain/depression]/extremely [anxiety/depression]); result: 5-digit health status profile that represents that person's level of reported problems on the five EQ-5D health dimensions
Stress: Perceived Stress (PSS-10) | week 0
  Perceived Stress Scale (PSS), Rating on a five-step scale from 1 (= never) to 5 (=very often), high stress is assumed from a total score of 20 points
Stress: Perceived Stress (PSS-10) | week 12
  Perceived Stress Scale (PSS), Rating on a five-step scale from 1 (= never) to 5 (=very often), high stress is assumed from a total score of 20 points
Stress: Perceived Stress (PSS-10) | week 36
  Perceived Stress Scale (PSS), Rating on a five-step scale from 1 (= never) to 5 (=very often), high stress is assumed from a total score of 20 points
Stress: Coping Strategies (CISS) | week 0
  Short version of the Coping Inventory for Stressful Situations (24 items); Rating on a five-step scale from 1 (= not at all) to 5 (= very much); sum score for each coping strategy; higher scores indicate a greater use of that particular coping strategy
Stress: Coping Strategies (CISS) | week 12
  Short version of the Coping Inventory for Stressful Situations (24 items); Rating on a five-step scale from 1 (= not at all) to 5 (= very much); sum score for each coping strategy; higher scores indicate a greater use of that particular coping strategy
Stress: Coping Strategies (CISS) | week 36
  Short version of the Coping Inventory for Stressful Situations (24 items); Rating on a five-step scale from 1 (= not at all) to 5 (= very much); sum score for each coping strategy; higher scores indicate a greater use of that particular coping strategy
Core Self-Evaluation by CSES | week 0
  Core Self-Evaluation (CSES), 12 items on five-point Likert scale, 1 indicates disagreement and 5 indicates full agreement. High scores on the CSES represents a positive, confident, and self-efficacious person
Core Self-Evaluation by CSES | week 12
  Core Self-Evaluation (CSES), 12 items on five-point Likert scale, 1 indicates disagreement and 5 indicates full agreement. High scores on the CSES represents a positive, confident, and self-efficacious person
Core Self-Evaluation by CSES | week 36
  Core Self-Evaluation (CSES), 12 items on five-point Likert scale, 1 indicates disagreement and 5 indicates full agreement. High scores on the CSES represents a positive, confident, and self-efficacious person
Utilization of medical services | week 0
  Number of visits
Utilization of medical services | week 12
  Number of visits
Utilization of medical services | week 36
  Number of visits
Days of work disability | week 0
  Number of days
Days of work disability | week 12
  Number of days
Days of work disability | week 36
  Number of days
Anxiety and depression by HADS | week 0
  Hospital Anxiety and Depression Scale (HADS), 14 items (7 each for depressive symptoms or symptoms of anxiety). The two summated scores of the summated scales HADS-A and HADS-D range between 0 and 21. high scores indicate depressivness and anxiety.
Anxiety and depression by HADS | week 12
  Hospital Anxiety and Depression Scale (HADS), 14 items (7 each for depressive symptoms or symptoms of anxiety). The two summated scores of the summated scales HADS-A and HADS-D range between 0 and 21. high scores indicate depressivness and anxiety.
Anxiety and depression by HADS | week 36
  Hospital Anxiety and Depression Scale (HADS), 14 items (7 each for depressive symptoms or symptoms of anxiety). The two summated scores of the summated scales HADS-A and HADS-D range between 0 and 21. high scores indicate depressivness and anxiety.
Qualitative Interviews | week 12
  Qualitative interviews for gaining further insights into patients experiences
Adverse events | week 12
  all adverse events
Adverse events | week 36
  all adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jost Langhorst, Prof. Dr., Principal Investigator — University of Duisburg-Essen/Sozialstiftung Bamberg
Locations (1):
- Sozialstiftung Bamberg, Bamberg, Bavaria, Germany